CLINICAL TRIAL: NCT00101751
Title: Efficacy and Safety of a Standard Titration Algorithm Coupled With a Conventional Dietary Intervention or Intensive Dietary Intervention Versus a Standard Titration Algorithm, Alone, in Patients With Type 2 Diabetes Initiating NovoLog® Mix 70/30 Therapy
Brief Title: INITIATE Plus (INITiation of Insulin to Reach A1c TargEt) Study
Acronym: INITIATE plus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-2192
Record Dates: First submitted 2005-01-12; First posted 2005-01-13 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: biphasic insulin aspart
Behavioral: dietary regimen

SUMMARY:
This trial is conducted in the United States of America (USA). The purpose of this study is to compare the effectiveness and safety of a biphasic insulin aspart standard titration regimen when coupled with dietary intervention to standard titration without dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4877 (Actual)
Dates: Start 2004-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
HbA1c and Incidence of hypoglycemia | After 24 weeks of treatment

SECONDARY OUTCOMES:
Postprandial glucose from 8-point SMBG spontaneously reported adverse events; any changes from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Clinical Trial Call Center, Princeton, New Jersey, United States

REFERENCES:
- [Derived] Trippe BS, Shepherd MD, Coulter FC, Bhargava A, Brett J, Chu PL, Oyer DS. Efficacy and safety of biphasic insulin aspart 70/30 in type 2 diabetes patients of different race or ethnicity (INITIATEplus trial). Curr Med Res Opin. 2012 Jul;28(7):1203-11. doi: 10.1185/03007995.2012.686444. Epub 2012 Jun 25. PMID 22509859
- [Derived] Oyer DS, Shepherd MD, Coulter FC, Bhargava A, Deluzio AJ, Chu PL, Trippe BS; Initiateplus Study Group. Efficacy and tolerability of self-titrated biphasic insulin aspart 70/30 in patients aged >65 years with type 2 diabetes: an exploratory post hoc subanalysis of the INITIATEplus trial. Clin Ther. 2011 Jul;33(7):874-83. doi: 10.1016/j.clinthera.2011.05.093. Epub 2011 Jul 8. PMID 21741089
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com